CLINICAL TRIAL: NCT00520000
Title: A Phase I Trial of Carboplatin and Abraxane in Patients With Solid Tumors
Brief Title: Carboplatin and Paclitaxel Albumin-Stabilized Nanoparticle Formulation in Treating Patients With Advanced or Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LCCC0412; CDR0000561620 (Other: PDQ number); NCT00254098 (obsolete NCT alias)
Record Dates: First submitted 2007-08-21; First posted 2007-08-23 (Estimated); Last update posted 2012-03-06 (Estimated); Status verified 2012-03

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Carboplatin; Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Weekly Arm (Active Comparator): Carboplatin day 1, abraxane days 1, 8, 15 every 28 day cycle
  Interventions: Drug: Carboplatin; Drug: Abraxane
- Every 3 week Arm (Experimental): Carboplatin day 1, abraxane day 1, every 21 day cycle
  Interventions: Drug: Carboplatin; Drug: Abraxane
- Arm C (Experimental): Carboplatin day 1, abraxane day 1, 8 every 21 day cycle
  Interventions: Drug: Carboplatin; Drug: Abraxane

INTERVENTIONS:
Drug: Carboplatin — standard dose of area under the curve (AUC) AUC of 6 in all arms
  Other Names: Paraplatin
Drug: Abraxane — 75mg/m2 - 150 mg/m2 given on days 1, 8, 15 of every 28 day cycle
  Other Names: Paclitaxil
  Arms: Weekly Arm
Drug: Abraxane — 180mg/m2 - 340mg/m2, repeated every 21 days
  Other Names: Paclitaxil
  Arms: Every 3 week Arm
Drug: Abraxane — 100mg/m2 - 175/mg/m2 given on days 1, 8 of every 21 day cycle
  Other Names: Paclitaxil
  Arms: Arm C

SUMMARY:
RATIONALE: Drugs used in chemotherapy such as paclitaxel albumin-stabilized nanoparticle formulation and carboplatin work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving paclitaxel albumin-stabilized nanoparticle formulation together with carboplatin may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects, the best way to give, and the best dose of paclitaxel albumin-stabilized nanoparticle formulation when given together with carboplatin in treating patients with advanced or metastatic solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose (MTD) of paclitaxel albumin-stabilized nanoparticle formulation given once weekly for 3 weeks when administered with carboplatin given once every 4 weeks.
* Determine the MTD of paclitaxel albumin-stabilized nanoparticle formulation given once every 3 weeks when administered with carboplatin given once every 3 weeks.
* Determine the MTD of paclitaxel albumin-stabilized nanoparticle formulation given in weeks 1 and 2 when administered with carboplatin given once every 3 weeks.
* Evaluate sequence-dependent effects on toxicity and pharmacokinetics in the combination of paclitaxel albumin-stabilized nanoparticle formulation and carboplatin.

Secondary

* Explore the antitumor activity of paclitaxel albumin-stabilized nanoparticle formulation given once weekly or once every 3 weeks.

OUTLINE: Patients are assigned to 1 of 3 treatment arms.

* Arm I: Patients receive carboplatin IV over 30 minutes on day 1 and paclitaxel albumin-stabilized nanoparticle formulation IV over 30 minutes on days 1, 8, and 15. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients receive carboplatin IV over 30 minutes on day 1 and paclitaxel albumin-stabilized nanoparticle formulation IV over 30 minutes on day 1. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
* Arm III: Patients receive carboplatin IV over 30 minutes on day 1 and paclitaxel albumin-stabilized nanoparticle formulation IV over 30 minutes on days 1 and 8. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

Patients in arms I and II undergo blood sample collection periodically for pharmacokinetic studies.

After completion of study treatment, patients are followed at 30 days.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

Inclusion criteria:

* Histologically or cytologically confirmed solid tumor

  * Advanced or metastatic disease
* Measurable or evaluable disease
* Must meet 1 of the following criteria:

  * Failed a standard therapy
  * Not a candidate for standard therapy
  * Have a disease for which there is no defined standard therapy

Exclusion criteria:

* Symptomatic brain metastases

PATIENT CHARACTERISTICS:

Inclusion criteria:

* ECOG performance status 0-2
* Life expectancy ≥ 8 weeks
* Absolute neutrophil count > 1,500/mm^3
* Platelet count > 100,000/mm^3
* Hemoglobin > 8.0 g/dL
* Total bilirubin normal
* Serum creatinine normal OR creatinine clearance ≥ 60 mL/min
* AST and ALT ≤ 2.5 x upper limit of normal
* Negative pregnancy test

Exclusion criteria:

* Pregnant or lactating
* Prior anaphylactic reaction or severe allergic reaction to paclitaxel and/or docetaxel
* Active infection that requires treatment with antibiotics for > 4 weeks
* Uncontrolled congestive heart failure
* Symptomatic coronary artery disease or heart block
* Myocardial infarction within the past 3 months
* Peripheral neuropathy ≥ grade 2 from any cause

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy, radiotherapy, or any other therapy for malignancy within the past 3 weeks
* No concurrent filgrastim, pegfilgrastim, or sargramostim during the first course of therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2004-12; Primary Completion 2006-05 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of Abraxane | 28 days
  To determine the maximum tolerated dose (MTD) of Abraxane weekly days 1, 8, 15 with a carboplatin dose of AUC=6 given on day 1 of a 28 day cycle
Maximum Tolerated Dose (MTD) of Abraxane given with Carboplatin | 21 days
  To determine the MTD of Abraxane given every 3 weeks with carboplatin given on day 1 of a 21 day cycle
Sequence-dependent toxicity | 28 days
  To determine if there is any correlation to toxicity based on the order Abraxane and carboplatin are adminstered

CONTACTS AND LOCATIONS:
Overall Officials: Thomas E. Stinchcombe, MD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center